CLINICAL TRIAL: NCT00405171
Title: Efavirenz to Nevirapine Switch in HIV-1 Infected Patients With Severe Dyslipidemia: A Randomized Controlled Study
Brief Title: Efavirenz to Nevirapine Switch and Low-Density Lipoprotein (LDL)-Dyslipidemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SIROCCO
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: HIV Infections; Hypercholesterolemia; Antiretroviral Therapy
Keywords: Efavirenz; Nevirapine; Dyslipidemia; HIV
MeSH Terms: conditions — HIV Infections; Hypercholesterolemia; Dyslipidemias | interventions — Nevirapine

INTERVENTIONS:
Drug: Nevirapine

SUMMARY:
Dyslipidemia and coronary heart disease (CHD) are increasingly recognized in persons with human immunodeficiency virus (HIV) infection. Many antiretrovirals, including efavirenz (EFV), are associated with increases in serum lipids. The investigators investigated whether stopping EFV and replace EFV by nevirapine can reduce significantly Low-Density Lipoprotein cholesterol, while keeping virologic control of HIV.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected adults, who were receiving antiretroviral therapy including efavirenz for at least 6 months
* plasma HIV RNA<400 cp/ml during the previous 4 months on 2 occasions 14 days apart
* Severe dyslipidemia with Low-Density Lipoprotein cholesterol (LDL-c) >3.4 mmol/L in the presence of at least one of the 3 following coronary heart disease (CHD) risk factors: age>45 among males or age>55 among females, hypertension, current smoking, family history of CHD
* Low-Density Lipoprotein cholesterol (LDL-c)>4.1 mmol/L regardless of CHD risk factors.

Exclusion Criteria:

* Protease inhibitors use within the previous 6 months,
* Prior exposure to nevirapine
* Asparate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5N if hepatitis virus B or C were negative
* AST or ALT>1.25N if hepatitis virus B or C were positive
* Fasting glycemia>1.26g/L,
* Current CHD
* Triglycerides>4.6 mmol/L
* Introduction of lipid lowering drugs, corticoïds, retinoïds and betablockers within the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-06; Study Completion 2006-02

PRIMARY OUTCOMES:
Decrease in LDL cholesterol between baseline and week 52

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Parienti, MD, Principal Investigator — University Hospital, Caen; Renaud Verdon, MD, PhD, Study Chair — Côte de Nacre
Locations (1):
- Côte de Nacre University hospital, Caen, France

REFERENCES:
- [Background] Parienti JJ, Peytavin G, Reliquet V, Verdon R, Coquerel A. Pharmacokinetics of the treatment switch from efavirenz to nevirapine. Clin Infect Dis. 2010 Jun 1;50(11):1547-8. doi: 10.1086/652718. No abstract available. PMID 20433360
- [Result] Parienti JJ, Massari V, Rey D, Poubeau P, Verdon R; SIROCCO study team. Efavirenz to nevirapine switch in HIV-1-infected patients with dyslipidemia: a randomized, controlled study. Clin Infect Dis. 2007 Jul 15;45(2):263-6. doi: 10.1086/518973. Epub 2007 Jun 6. PMID 17578790